CLINICAL TRIAL: NCT04596410
Title: Double-blind, Randomized, Multi-center, Non-inferiority Clinical Trial Comparing Two Photobiomodulation Protocols in the Analgesia of Chemotherapy-induced Oral Mucositis in Children
Brief Title: Photobiomodulation Protocols in the Analgesia of Chemotherapy-induced Oral Mucositis in Children
Acronym: CURALASE01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC31/19/0556
Record Dates: First submitted 2020-09-04; First posted 2020-10-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Mucositis Oral
Keywords: Children; Oral mucositis; Chemotherapy; Photobiomodulation
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT applied every other day (Experimental): Low-level laser therapy (LLLT) protocol combining red and infrared wavelengths applied every other day
  Interventions: Radiation: LLLT applied every other day
- LLLT applied daily (Active Comparator): Low-level laser therapy (LLLT) protocol combining red and infrared wavelengths applied every day
  Interventions: Radiation: LLLT applied daily

INTERVENTIONS:
Radiation: LLLT applied every other day — Low-level laser therapy (LLLT) protocol combining red and infrared wavelengths applied every other day
  Arms: LLLT applied every other day
Radiation: LLLT applied daily — Low-level laser therapy (LLLT) protocol combining red and infrared wavelengths applied daily
  Arms: LLLT applied daily

SUMMARY:
Chemotherapy-induced oropharyngeal mucositis (OM) negatively impacts the quality of life of adult and pediatric patients by causing pain, dysphagia, dysgeusia and dysphonia.

Photobiomodulation (PBM) by low level laser therapy (LLLT), light therapy of low level of red and infrared wavelengths (630-1000 nm) has been recommended since 2014 in patients treated with high-dose chemotherapy for bone marrow transplantation. Available pediatric studies highlighted positive/promising results of PBM with excellent safety and no adverse effects. Nevertheless, a wide variety of application parameters is described in the literature, with no consensus guidelines.

Considering the lack of standardized protocol of photobiomodulation in the pediatric population as well as the burden and cost of a daily application, investigators have decided to conduct, for the first time in children of 3 years of age or older, a multicenter, randomized, double-blind, non-inferiority clinical trial to compare two PBM protocols with same PBM parameters, combining red and infrared wavelengths, but with different frequencies of laser application (daily versus every other day), in the treatment of chemotherapy-induced OM of WHO grade 2 or higher.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children aged ≥ 3 years and < 18 years.
2. Hospitalization in an oncology or hematology department in the participating centres.
3. Patients with oropharyngeal mucositis of grade 2 or higher (WHO grading system) related to cancer chemotherapy, including conditioning for Hematopoietic Stem Cell Transplantation (HSCT).
4. Written informed consent of both patient's holders of parental authority, and patient's assent when applicable.
5. Patients affiliated to a French Social Security insurance or equivalent social protection.
6. Absence of any physical or psychological disability that may interfere with the LLLT application.

Exclusion Criteria:

1. Patients with a solid cancer lesion in the area of low-level laser application.
2. History of cervicofacial radiotherapy.
3. Application of low-level laser therapy for oral mucositis within 2 weeks prior to randomization.
4. Hyperthyroidism defined by TSH < 0.4 IU/mL at inclusion.
5. Patients susceptible to epilepsy seizure.
6. Patients with pacemaker.
7. Patients refusing to wear retinal goggles during low-level laser 1. Patients with a solid cancer lesion in the area of low-level laser application.
8. Patients protected by law (guardianship and safeguarding of justice).
9. Pregnant female patients as determined by positive serum pregnancy test at screening.
10. Lactating female patients who are actively breast feeding.
11. Participation in another clinical trial involving oral care.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 406 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Session evaluation | Throught treatment period up to 1 month
  Duration (in days) from the day of first PBM session up to the day of first measurement when patient has no longer WHO grade 2 or higher chemotherapy-induced OM related pain at 2 consecutive measurements before the next scheduled PBM session (either active laser application or matching placebo application)

SECONDARY OUTCOMES:
Production costs evaluation | 2 months
  Production costs from the hospital perspective and efficacy (i.e. number of days after which a child has no longer mucositis related pain as described in the primary endpoint section) to build Incremental Cost-Effectiveness Ratio (ICER) comparing every other day LLLT application versus with daily LLLT application.
Health insurance evaluation | 2 months
  Costs of inpatient hospital stays from the French health insurance perspective.
OM duration evaluation | Throught treatment period up to 1 month
  Duration (in days) of chemotherapy-induced OM of WHO grade 2 or higher between the day of first PBM session up to the day of first measurement when patient has no longer WHO grade 2 or higher chemotherapy-induced OM at 2 consecutive measurements before the next scheduled PBM session (either every other day application or daily application).
OM occurrence | 2 months
  Occurrence of chemotherapy-induced OM of WHO grade 3 or 4 (deterioration of the clinical situation).
Feed evaluation | 2 months
  Occurrence of enteral feeding.
Analgesic consumption | 2 months
  Duration (in days) of consumption of step 2 and step 3 analgesics during chemotherapy-induced OM of WHO grade 2 or higher.
PBM evaluation | Through treatment period up to 1 month
  Duration (in days) from the day of first PBM session up to the day of first measurement when patient has no longer WHO grade 2 or higher chemotherapy-induced OM related pain at 2 consecutive measurements before the next scheduled PBM session (either active laser application or matching placebo application) as evaluated, regardless of patient's age, with the ChIMES scale and use of step 3 analgesics.
Pain change evaluation | From baseline to each day of PBM session
  Change over time in WHO grade 2 or higher chemotherapy-induced OM related pain, as assessed by pain scales (HEDEN (Hétero Evaluation Douleur Enfant) mucositis scale (5 items ranging from 0 to 2) or VAS (ranging from 0 to 10)depending on patient's age category, and Children's International Mucositis Evaluation Scale (4 items ranging from 0 to 5) whatever patient's age category)
Adverse events occurrence | 2 months
  Occurrence of adverse events reported according to descriptions and grading scale found in NCI CTCAE version 5.0.
thyroid-stimulating hormone (TSH) evolution | From baseline to 2 months
  TSH shift from baseline value classified according to the following three categories: "< 0.4 IU/mL", "[0.4 - 10] IU/mL", "> 10 IU/mL", to value at D14-31 after end of WHO grade 2 or higher chemotherapy-induced OM classified according to the same three categories.

CONTACTS AND LOCATIONS:
Overall Officials: Marlène PASQUET, Principal Investigator — University Hospital, Toulouse
Locations (16):
- France (16):
  - University hospital of Toulouse, Toulouse, Occitanie
  - University hospital of Angers, Angers
  - University hospital of Besançon, Besançon
  - University hospital of Grenoble, Grenoble
  - University hospital of Lille, Lille
  - University hospital of Limoges, Limoges
  - Hôpital La Timone, Marseille
  - University hospital of Nancy, Nancy
  - University Hospital of Nice, Nice
  - Armand Trousseau Hospital, Paris
  - University hospital of Poitiers, Poitiers
  - University hospital of Reims, Reims
  - University hospital of Rouen, Rouen
  - University hospital of Saint-Etienne, Saint-Etienne
  - University hospital of Strasbourg, Strasbourg
  - University Hospital of Tours, Tours